CLINICAL TRIAL: NCT06834295
Title: An Open-label, Single-dose Study To Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]Vapendavir in Healthy Male Subjects
Brief Title: A Study to Evaluate Metabolism, Excretion, and Mass Balance of [14C]Vapendavir
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Altesa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALT VPV-102
Record Dates: First submitted 2025-02-11; First posted 2025-02-19 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy Males
Keywords: ADME Study in Healthy Males

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label, non-randomized, single-dose of [14C]Vapendavir (Experimental): Single oral dose of [14C]Vapendavir
  Interventions: Drug: Vapendavir

INTERVENTIONS:
Drug: Vapendavir — Single oral dose of [14C]vapendavir

SUMMARY:
The goal of this clinical trial is to assess how the body processes, breaks down and removes a new test medicine (vapendavir) from the body in healthy male participants.The main question it aims to answer is how the body handles the test medicine. In order to do that, the test medicine will be radiolabeled to track the test medicine in the body.

Healthy male participants who meet entry criteria will be admitted to the clinic for a duration of approximately 9 days (Day -1 to Day 8). Participants will be admitted in the evening on the day before dosing (Day -1). Participants will take a single oral dose of radiolabeled vapendavir on Day 1 and have samples collected and safety tests completed during various times throughout their stay in the the clinic. The safety tests will provide additional information on the safety and tolerability of the test medicine.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent
* Must be willing and able to communicate and participate in the whole study
* Participants must demonstrate their ability to swallow 8 capsules
* Aged 30 to 65 years inclusive at the time of signing informed consent
* Must agree to adhere to the study contraception requirements
* Healthy male participants according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs, 12- lead ECG, and laboratory safety tests without any clinically significant abnormalities
* Body mass index (BMI) of 18.0 to 35.0 kg/m2 as measured at screening
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
* Acute diarrhea or constipation in the 7 days before the predicted Day 1
* Participants who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Clinically significant abnormal laboratory values at screening as judged by the investigator
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results
* Evidence of renal impairment at screening
* Participants who have received any IMP in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
* Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 3 g of paracetamol per day) in the 14 days before dosing
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week (1 unit = 1⁄2 pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 = 125 mL glass of wine, depending on type)
* A confirmed positive alcohol breath test
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes or nicotine replacement products and those who have used these products within the last 12 months
* A confirmed breath carbon monoxide reading of greater than 10 ppm
* Confirmed positive drugs of abuse test result
* Male participants with pregnant or lactating partners
* Participants who are, or are immediate family members of, a study site or sponsor or employee
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male subjects
Enrollment: 8 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
To determine the mass balance recovery after a single oral dose of carbon-14 ([14C])vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Mass balance recovery of total radioactivity in all excreta (urine and feces): CumAe and Cum%Ae.

SECONDARY OUTCOMES:
To determine the routes and rates of elimination of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Determination of routes and rates of elimination of [14C]vapendavir by Ae, %Ae, CumAe and Cum%Ae by interval.
To perform metabolite profiling and structural identification from plasma, urine and fecal samples. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Identification of the chemical structure of each metabolite accounting for greater than or equal to 10% of circulating radioactivity in plasma ("AUC pool"), and accounting for greater than or equal to 10% of the dose in urine (from urine pools) and feces (fecal homogenate pools) will be performed.
To identify the chemical structure of each metabolite accounting for more than 10% of circulating total radioactivity or accounting for 10% or more of the dose in excreta. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Identification of the chemical structure of each metabolite accounting for more than 10% by AUC of circulating total radioactivity or accounting for 10% or more of the dose in excreta.
To evaluate the extent of distribution of total radioactivity into blood cells. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Evaluation of whole blood: plasma concentration ratios for total radioactivity.
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Time prior to the first measurable concentration (Tlag)
To provide additional safety and tolerability information for vapendavir by assessing: incidence of adverse events (AEs), new physical examination findings and change from baseline for vital signs, electrocardiograms (ECGs), and laboratory safety tests. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Descriptive summaries for all safety data (AEs, vital signs, ECGs and safety laboratory assessments) will be provided.
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Time of maximum observed concentration (Tmax)
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Maximum observed concentration (Cmax)
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Area under the curve from time 0 to the time of last measurable concentration (AUC (0-last))
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Area under the curve from time 0 extrapolated to infinity (AUC (0-inf))
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Terminal elimination half-life (T1/2)
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  First order rate constant associated with the terminal (log-linear) portion of the curve (Ke)
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F)
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the cure extrapolated to infinity (AUCextrap)
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Mean residence time from time 0 to time of the last measurable concentration (MRT(0-last))
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days)
  Mean residence time from time 0 to extrapolated to infinity (MRT(0-inf))
To further explore the oral pharmacokinetic (PK) of vapendavir. To characterise the PK of vapendavir and total radioactivity in plasma following a single oral dose of [14C]vapendavir. | From enrollment until the mass balance criteria have been met (~ 8 days).
  Apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vd/F).

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided